CLINICAL TRIAL: NCT02985671
Title: National Clinical Study, Phase III, Multicenter, Randomized, Double-blind, Controlled, Parallel, to Evaluate the Superiority of the Fixed Association (Orfenadrine 35mg, Acetaminophen 325mg, Caffeine 65mg and Diclofenac Sodium 50mg) Compared to the Drug Comparator Voltaren® (Diclofenac Sodium 50mg), in the Treatment of Acute Episode of Mechanical Postural Low Back Pain.
Brief Title: To Evaluate the Superiority of Fixed Combination (Orfenadrine 35mg, Acetaminophen 325mg, Caffeine 65mg and Diclofenac Sodium 50mg) Compared to Voltaren® (Diclofenac Sodium 50mg) in the Treatment of Acute Postural Low Back Pain.
Acronym: Eiffel
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACH-TND-03(12/14)
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Postural Low Back Pain; Mechanical Low Back Pain
Keywords: Postural Low Back Pain; Mechanical Low Back Pain; Low Back Pain; acetaminophen; caffeine; orphenadrine; diclofenac sodium
MeSH Terms: conditions — Low Back Pain | interventions — Orphenadrine; Acetaminophen; Caffeine; Diclofenac; Drugs, Investigational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Drug & Voltaren Placebo (Experimental): Orphenadrine + acetaminophen + caffeine + diclofenac sodium & Placebo of Voltaren
  01 tablet of experimental drug (orphenadrine 35mg, acetaminophen 325mg, caffeine 65mg and diclofenac sodium 50mg) + 01 tablet of placebo of Voltaren, to be administrated orally, three times a day, respecting the interval of 08 hours between administrations, during 7 days.
  Interventions: Drug: orphenadrine, acetaminophen, caffeine and diclofenac sodium; Drug: Placebo (for Voltaren)
- Voltaren® + Experimental Drug Placebo (Active Comparator): Voltaren & Placebo of Orphenadrine + acetaminophen + caffeine + diclofenac sodium
  01 tablet of Voltaren + 01 tablet of placebo of experimental drug (orphenadrine, acetaminophen, caffeine and diclofenac sodium), to be administrated orally, three times a day, respecting the interval of 08 hours between administrations, during 7 days.
  Interventions: Drug: Diclofenac Sodium 50 MG; Drug: Placebo (for experimental drug)

INTERVENTIONS:
Drug: orphenadrine, acetaminophen, caffeine and diclofenac sodium — orphenadrine 35mg, acetaminophen 325mg, caffeine 65mg and diclofenac sodium 50mg tablet
  Other Names: experimental drug
  Arms: Experimental Drug & Voltaren Placebo
Drug: Diclofenac Sodium 50 MG — Voltaren (diclofenac sodium 50mg) tablet
  Other Names: active comparator; Voltaren
  Arms: Voltaren® + Experimental Drug Placebo
Drug: Placebo (for experimental drug) — tablet without active substances, manufactured to mimic experimental product tablet
  Other Names: Placebo (for orphenadrine + acetaminophen + caffeine + diclofenac sodium)
  Arms: Voltaren® + Experimental Drug Placebo
Drug: Placebo (for Voltaren) — tablet without active substances, manufactured to mimic Voltaren 50mg tablet
  Other Names: Placebo (for Voltaren 50mg)
  Arms: Experimental Drug & Voltaren Placebo

SUMMARY:
The purpose of this study is to determine whether the fixed combination of orphenadrine, acetaminophen, caffeine and diclofenac sodium is more effective in the treatment of an acute episode of mechanical postural low back pain than Voltaren®. Will be randomized 110 participants of both sexes, aged 18 years or older and less than 65 years of age with an acute episode of mechanical postural low back pain and they will be allocated to one of two treatment groups: Group 1: Fixed combination of orphenadrine, acetaminophen, caffeine and diclofenac sodium; or Group 2: Voltaren®

DETAILED DESCRIPTION:
The fixed combination of orphenadrine 35mg, acetaminophen 325mg, caffeine 65mg and diclofenac sodium 50mg aims to provide patients with anti-inflammatory, analgesic and myorelaxant action with adequate safety and tolerability profile.

Diclofenac is a nonsteroidal anti-inflammatory with analgesic, anti-inflammatory and antipyretic action and is effective in the treatment of a variety of acute and chronic inflammatory and painful conditions. Its anti-inflammatory effect occurs by inhibiting the synthesis of prostaglandins by inhibiting COX-1 and COX-2 in an equipotent manner.

Orphenadrine, on the other hand, is a central acting muscle relaxant that has analgesic and anticholinergic effects. It presents clinical efficacy in the treatment of painful conditions associated to pictures such as strains and sprains, especially of acute character, among other musculoskeletal conditions that present with pain and muscular contracture.

Concerning acetaminophen, its a drug with analgesic and antipyretic action as well as anti-inflammatory properties. It is widely used in a wide variety of pathologies with a focus on the treatment of mild to moderate pain. It is a non-opioid analgesic with action in the inhibition of cyclooxygenase and consequently in the production of prostaglandins, with potency similar to that of aspirin. It is the analgesic of choice for children, the elderly and pregnant women. It has been used successfully in the treatment of back pain. The association between acetaminophen and orphenadrine is known and clinically effective in analgesia, as well as the combination of acetaminophen and diclofenac, which also provides clinical efficacy in the management of acute postoperative pain.

Lastly, caffeine, an alkaloid belonging to the group of methylxanthines, is an agonist that competes with adenosine receptors, acting in these receptors in very varied areas, such as throughout the peripheral circulation and in the cerebral cortex. Caffeine enhances the effects of other analgesics, improves acetaminophen pharmacokinetics, and induces mood changes. All these mechanisms may contribute to improve the analgesic action of acetaminophen.

The association of non-steroidal anti-inflammatory, muscle relaxant, analgesic and caffeine in the symptomatic treatment of painful conditions associated with the musculoskeletal system is quite old.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and consent their participation in this clinical study, expressed by signing the Informed Consent Form (ICF);
2. Patient with acute low back pain who responds to the pain period less than or equal to 3 days and the minimum value of 40 mm in the VAS;
3. Research participants who perform simple RX of lumbosacral spine, with results within the limits of normality for the age group.

Exclusion Criteria:

1. Use of illicit drugs;
2. Fertile women who have had a positive pregnancy test in the urine or during gestation or breastfeeding;
3. Participants who present with allergic reaction, asthma or urticaria in response to exposure to aspirin, sulfonamides and other NSAIDs;
4. Women who do not agree to use acceptable contraceptive methods (oral contraceptive, intravenous contraceptive, intrauterine device (IUD), hormonal implant, barrier methods, hormonal transdermal patch and tubal ligation); except for those surgically sterile (bilateral oophorectomy or hysterectomy), menopause for at least one year, and participants who report not engaging in sexual practices or non-reproductive practices;
5. Participants with inflammatory conditions such as any rheumatic condition known as rheumatoid arthritis, osteoarthrosis (grade II, III and IV criteria of Kellgren and Lawrence, Annex IV), ankylosing spondylitis or psoriatic arthritis, chronic pain condition (greater than six weeks), primary or secondary neoplasia, moderate to severe scoliosis (greater than 40º), low back pain as a result of trauma, visceral disorder such as dysmenorrhea or endometriosis;
6. Known hypersensitivity to the components of the medicines used during the study;
7. Research participants who have had bacterial infection recently (last 90 days), affecting the spine, pelvic or abdominal region; as well as participants with a history of bacterial infection that affected the spine in a chronic way;
8. Research participants previously diagnosed with herniated disc, osteoid osteoma, arthroscopic narrowing of the spinal canal, spondyloarthropathies, spondylodiscites, renal calculus, calculitic cholecystitis, endometriosis, prostatitis, abdominal aortic aneurysm, chronic pelvic pain, pyelonephritis, perirenal abscesses and pancreatitis , rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia rheumatica, gout, episodes of acute monoarthritis compatible with pseudogout, Paget's disease, septic arthritis, avascular necrosis, Wilson's disease, hemochromatosis, alkaptonuria, primary osteochondromatosis, iritis, colitis, urethritis and skin rash;
9. Participants who present suspected or previous history of esophageal, gastric or duodenal ulcers, or bleeding before the first dose of study medication;
10. Research participants presenting with any chronic uncontrolled disease, such as diabetes, hypertension, chronic hepatic or renal disorders, or any clinical condition that, in the opinion of the investigator, may interfere with the study drug;
11. Participants presenting with inflammatory bowel disorders (eg, Crohn's disease or ulcerative colitis), significant coagulation defect or history of cardiovascular disease that may prevent the use of NSAIDs, such as congestive heart failure;
12. Any finding of clinical observation (clinical / physical assessment) that is interpreted by the investigating physician as a risk to the participation of the research participant in the clinical study;
13. History of lumbar spine surgery, of any nature;
14. Failure to understand and respond to the Roland Morris questionnaire, SF-36 quality of life questionnaire, and Participant's diary, and who do not have an accompanying person to assist him / her;
15. Participant with a history of malignant disease without documentation of remission / cure, eg, melanoma, leukemia, lymphoma, myeloproliferative diseases and renal cell carcinoma of any duration should be excluded;
16. Immunosuppressed participants;
17. Research participants who perform treatment for osteoporosis;
18. Diagnosis of equine cauda syndrome and / or acute severe neurological deficit (presence of motor or sensory changes in the lower limbs and positive Lasegue signal> 60o). Sphincter and anesthesia changes in saddle;
19. History of intense pain at minimal effort, progressive pain and night and persistent restriction of movement;
20. Research participants with unexplained weight loss (more than 10kg in three months);
21. Research participants who are performing some type of oral, physical or topical treatment for low back pain (eg acupuncture, local heat and yoga) and / or initiation of physiotherapy program in the last 2 months before the start of the study;
22. Participant in research that has participated in clinical study protocols in the last 12 (twelve) months (CNS Resolution 251, August 7, 1997, item III, subitem J), unless the investigator deems that there may be direct benefit To the same;
23. Use of prohibited drugs specified in item 11.2 of this protocol. If the participant makes use of acetylsalicylic acid, used as antiplatelet agent, the maximum dose of 200mg will be allowed;
24. Participant who has a relationship of kinship to second degree or bond with employees or employees of Sponsor and Research Center.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Superiority of the fixed association of orfenadrine 35 mg, acetaminophen 325 mg, caffeine 65 mg and diclofenac sodium 50 mg, compared to Voltaren® in the treatment of the acute mechanical postural low back pain. | 72 hours (± 7 hours) after initiation of treatment.
  The primary efficacy variable was the absolute variation of pain intensity measured by the EVA - Visual Analogue Scale of 100mm (0mm = no pain and 100mm = maximum pain) in relation to Baseline (V0), defined as EVA72-0 = (EVA72 - EVA0).

SECONDARY OUTCOMES:
Relief of pain in the treatment of acute postural mechanical low back pain throughout treatment. | 15', 30', 45', 60', 90', 120', 72h (±7h) and 168h (+48h) after the first administration of the drug for which the study participant was randomized.
  Absolute variation of pain intensity measured by EVA - Visual Analog Scale of 100mm (0mm = no pain and 100mm = maximum pain) in relation to the basal (V0).
Intensity of pain in the treatment of acute postural mechanical low back pain throughout treatment. | 24 hours and 48 hours after the first administration of the drug for which the study participant was randomized
  pain intensity measured by EVA - Visual Analog Scale of 100mm (0mm = no pain and 100mm = maximum pain) and reported daily in 24 and 48 hours after the first administration of the drug
Need for rescue medication to control acute pain between treatment groups during the study period. | 07 days
  Proportion of participants who needed at least one rescue medication during the study in each treatment group.
Number of rescue medication tablets used daily by the research participant in each treatment group. | 07 days
  Number of rescue medication tablets used daily by the baseline visit participant up to the final study visit in each treatment group as assessed by the research participant's diary.
Evaluation of the functional incapacity of the research participants. | 07 days
  Absolute variation of the total score of the Roland-Morris functional disability questionnaire assessed at visits V1 and VF, in relation to the total baseline score (V0). This questionnaire consists of 24 dichotomous items (0 = No and 1 = Yes) and thus the total score ranges from 0 to 24 points (0 = no complaints and 24 = very serious limitations).
Evaluation of the quality of life of the research participants. | 07 days
  Absolute variation of the score of each SF-36 quality of life questionnaire domain (functional capacity, limitation for physical aspects, pain, general health status, vitality, social aspects, emotional aspects and mental health) evaluated in the final visit (VF), in relation to the basal score (V0). The result of each domain of this questionnaire ranges from 0 to 100 points (0 = worst state and 100 = best state).
Evaluation of participant satisfaction with treatment. | 07 days
  Satisfaction of the research participant with the treatment, evaluated in the final visit (VF) by means of the visual analog scale of 100 points (EVA of 100mm, being 0mm = totally unsatisfied and 100mm = totally satisfied).
Assess the safety of treatments during the study period. | The first dose of the study drug up to 30 days after the end of treatment.
  Incidence of adverse events (AEs) recorded from the first dose of the study drug up to 30 days after the end of treatment, but all adverse events occurring after the signing of the ICF will be collected and reported.
Assess the safety of treatments during the study period. | Day of V1 and day of VF.
  Absolute variation of the vital signs measured in visits V1 and VF in relation to the baseline visit (V0).
Assess the safety of treatments during the study period. | Day of V1 and day of VF.
  Proportion of participants with clinical or physical changes, considered relevant according to the researcher's criteria, at visits V1 and VF in relation to the baseline visit (V0).
Assess the safety of treatments during the study period. | Day of V0 and day of VF.
  Proportion of participants with altered laboratory tests, considered clinically relevant according to the researcher's criteria, at the baseline visit (V0) and at the final visit (VF) of the study.
Assess the safety of treatments during the study period. | Day of V0.
  Proportion of participants with alterations in the ECG exam, considered clinically relevant according to the researcher's criteria, observed in visits V0.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro C Junior, M.D., Principal Investigator — Allergisa Search Dermato Cosmetic Ltda.; Morton A Scheinberg, M.D., Principal Investigator — AACD - Association of Assistance to the Disabled Child; Pedro Henrique I Pohl, M.D., Principal Investigator — Center for Multidisciplinary Studies CEPES; Pérola G Plapler, M.D., Principal Investigator — Clinical Research Center IOT HCFMUSP; Suely S Roizenblatt, Principal Investigator — CDEC Brazil - Center for the Development of Clinical Studies Brazil

IPD SHARING:
Plan to Share IPD: No